CLINICAL TRIAL: NCT02677662
Title: Longitudinal Acute Air Pollution Systemic Effects (LAPSE)
Brief Title: Longitudinal Acute Air Pollution Systemic Effects
Acronym: LAPSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, Jenny Bosson, MD, PhD, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015-69-31M
Record Dates: First submitted 2016-01-21; First posted 2016-02-09 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Diesel exhaust; Oxidative stress; Systemic inflammation; Air pollution
MeSH Terms: interventions — Vehicle Emissions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filtered air exposure (Sham Comparator): 2 hour exposure to filtered air during intermittent exercise or rest.
  Interventions: Other: Filtered air
- Diesel exhaust exposure (Experimental): 2 hour exposure to dilute diesel exhaust (approximate PM10 (particulate matter<10um) concentration 300 mcg/m3) during intermittent exercise or rest.
  Interventions: Other: Diesel Exhaust

INTERVENTIONS:
Other: Diesel Exhaust — Dilute diesel exhaust
  Arms: Diesel exhaust exposure
Other: Filtered air — Filtered air
  Arms: Filtered air exposure

SUMMARY:
Air pollution continues to be a key global issue with many governments focusing great attention on air quality legislation because of its harmful environmental and health impacts. Whilst there is much that remains unknown about the mechanisms underlying the negative health effects of air pollution, it is generally acknowledged that air pollution exposure leads to an increase in cardiovascular, cerebrovascular and respiratory mortality and morbidity. The current study will investigate systemic effects during a 72 hour period after a controlled diesel exhaust exposure.

DETAILED DESCRIPTION:
Exposure to air pollution (both indoor and outdoor sources) contributes to the premature deaths of 7 million people each year, primarily linked to cardiovascular and respiratory conditions. Within the complex mixture which air pollution comprises, combustion derived particulate matter (PM) has been suggested as one of the most harmful components to the cardiopulmonary system. In urban areas PM derived from combustion originates largely from diesel vehicles.

Numerous experimental chamber studies have demonstrated respiratory as well as cardiovascular dysfunctions after the inhalation of diesel exhaust. Many of these dysfunctions are driven by inflammation and oxidative stress. There is much less knowledge concerning the systemic effects of diesel exhaust exposure, and especially over longer time courses than 24 hours.

The investigators aim to investigate the time course of systemic effects (such as markers of inflammation, cardiovascular dysfunction, and oxidative stress) in blood and urine samples taken after a diesel exhaust exposure. The effects of exercise or rest in an experimental chamber exposure will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Normal clinical examination
* Normal EKG
* Normal routine blood tests
* Normal lung function
* Normal skinprick test

Exclusion Criteria:

* Cardiovascular disease
* Diabetes Mellitus
* Asthma and/or allergy
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers | 72 hours
  In blood samples (total and differential counts

SECONDARY OUTCOMES:
Oxidative stress markers | 72 hours
  In blood samples (ox-LDL, ROS)
Cardiovascular biomarkers | 72 hours
  In blood samples (sTM, hsCRP, syndecan-1)
Metabolomics | 72 hours
  Mass spectrometry based metabolomics in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Bosson, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided